CLINICAL TRIAL: NCT03739567
Title: Postoperative Pain in Children Aged From 3 to 5 Years Following Full Mouth Dental Rehabilitation Under General Anesthesia
Brief Title: Postoperative Pain in Children Aged From 3 to 5 Years Following Full Mouth Dental Rehabilitation Under General Anesthesia. A Cross-sectional Study. Rehabilitation Under General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mostafa Ahmed, Master student in Cairo university, Cairo University
Other Study IDs: CEBD-CU-2018-11-08
Record Dates: First submitted 2018-11-07; First posted 2018-11-14 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-11

CONDITIONS: Post-operative Pain
Keywords: General anesthesia, clinical manifestations. .
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the purpose of this study is monitoring Postoperative pain in Children Aged from 3 to 5 years following Full mouth Dental Rehabilitation under General Anesthesia

DETAILED DESCRIPTION:
The study's investigators will record all data related to the immediate postoperative period during the child's stay in the post anesthetic recovery room (PAR).

Just prior to discharge home, the child's discomfort will be measured using Face, Legs, Activity, Cry, and Consolability Pain Assessment Tool (FLACC).

Postoperative data is collected by the same investigator who contacted caregivers by phone at 4 postoperative times: 1, 3, 7, and 30 days after the DRGA using The Dental Questionnaire.

When a participant cannot be reached on the scheduled day, the information is collected on the nearest subsequent day.

The postoperative assessment included: the questioner and an inquiry about the use of medications; the child's ability to eat a regular diet; and "mouth-related" complaints other than dental discomfort.

Dental discomfort is assessed in this study by 2 scales:

the FLACC (Table 1) and The Dental Questioner (Table 2).

FLACC pain assessment tool. The FLACC scale was originally developed to quantify postoperative pain in infants from 2 months old to children up to 7-years-old.(7) This scale assesses 5 aspects of behavior: (F) facial expression; (L) leg movement; (A) activity; (C) cry; and (C) consolability. The range for the total score is from 0 (no pain) to 10 (intense pain). The examiner is standardized to use of the FLACC by a PAR nurse who was experienced in scoring pain with this scale.

The Dental Questioner. The questionnaire covered the following items: did the Child have pain, bleeding from dental origin, sore throat, fever, vomiting, inability to eat, sleepiness, drowsiness, cough, nausea or psychological changes?

ELIGIBILITY:
Inclusion Criteria:

* Egyptian dental children undergoing full mouth dental rehabilitation under general anesthesia (3-5 years old )
* Children selected from pediatric dentistry and dental public health department Faculty of dentistry Cairo University
* Children with no developmental delay.
* Children with normal physical status.
* Parents who can be communicated well

Exclusion Criteria:

* Parents refusing participation in the study.
* Parents who cannot be communicated well
* Children with developmental abnormalities

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children attending the outpatients' clinic of pediatric Dentistry and Public Health Faculty of Dentistry Cairo University-Egypt in the period of three months. (With average 30 patients in week ).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Dental Discomfort Questionnaire | 3 monthes
  Numerical Rating Pain Scale (Outcome measuring device)

CONTACTS AND LOCATIONS:
Overall Officials: Amr ezzat, professor, Study Director — Cairo University